CLINICAL TRIAL: NCT01865409
Title: Does Kangaroo Care Effects on Heart Rate Variability in Neonates
Brief Title: Effect of Kangaroo Care on Heart Rate Variability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fatih University (Other)
Responsible Party: Principal Investigator, Mehmet Kenan Kanburoglu, MD Kanburoglu, neonatologist, Fatih University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B 30 FTH 0 20 00 00 / 1503
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Immaturity; Oral Intolerance; Postnatal Adaptation
Keywords: Newborn; Prematures; Feeding difficulty; Kangaroo Care; Heart rate variability
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kangoroo care (Active Comparator): While performing "Kangaroo care" the infant should be held skin-to-skin contact with her mother for 30-60 minutes. The baby, who is naked except for a diaper and a piece of cloth covering his or her back (either a receiving blanket or the parent's clothing), is placed in an upright position against a parent's bare chest. The values of heart rate variability will be measured during and also without Kangaroo Care in the same infants but different times.
  Interventions: Behavioral: Kangaroo Care

INTERVENTIONS:
Behavioral: Kangaroo Care — Kangaroo care is a technique practiced on newborn, usually preterm, infants wherein the infant is held, skin-to-skin, with an adult.
  Other Names: Kangaroo Mother Care; Skin to skin contact

SUMMARY:
Physiological processes leading to a preterm infant to be able to feed orally has not been fully understood. The investigators hypothesized that maturation of autonomic nervous system may play a major role in this process and kangaroo care may accelerate this maturation. The investigators will use heart rate variability to measure the maturation of autonomic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants between 32 t0 35 weeks old
* After 7 days of extra-uterine life

Exclusion Criteria:

* Sepsis, infection
* Cardiac disease
* Intraventricular hemorrhage, patent ductus arteriosus, necrotizing enterocolitis

Ages: 32 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
HRV-Sympathetic-Short Measurement-LF | 5 Minutes
  By using Holter monitorization for 24 haur. LF (frequency domain, low frequency measurement): The low-frequency (LF) spectra represents predominantly sympathetic with some parasympathetic influence in the 0.04-to-0.15 Hz range.

SECONDARY OUTCOMES:
Time Domain Measurements of HRV | 5 Minutes
  By using Holter monitorization for 24 haur, 5 different measurements get by 5 minutes heart rate analysis: SDNN, SDANN,SDNN index,Rmssd,pNN50 SDNN: ms, Standard deviation of all NN intervals. SDANN: ms Standard deviation of the averages of NN intervals in all 5 min segments of the entire recording.
  SDNN index: ms, mean of the standard deviations of all NN intervals for all 5 min segments of the entire recording RMSSD: ms, The square root of the mean of the sum of the squares of diVerences between adjacent NN intervals.
  pNN50: % NN50 count divided by the total number of all NN intervals

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kenan Kanburoglu, MD, Study Director — Neonatologist; Mehmet Nevzat Cizmeci, MD, Principal Investigator — Neonatologist; Mustafa Mansur Tatli, MD, Prof, Study Chair — Neonatologist
Locations (1):
- Fatih University School of Medicine, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Srinivasan L, Harris MC. New technologies for the rapid diagnosis of neonatal sepsis. Curr Opin Pediatr. 2012 Apr;24(2):165-71. doi: 10.1097/MOP.0b013e3283504df3. PMID 22273634
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Harrison TM. Trajectories of parasympathetic nervous system function before, during, and after feeding in infants with transposition of the great arteries. Nurs Res. 2011 May-Jun;60(3 Suppl):S15-27. doi: 10.1097/NNR.0b013e31821600b1. PMID 21543958